CLINICAL TRIAL: NCT07369193
Title: Immersive AOT: Multisensory Stimulation and Neurophysiological Correlates - A Pilot Study
Brief Title: Immersive AOT: Multisensory Stimulation and Neurophysiological Correlates in Children With Cerebral Palsy and Typical Development - A Pilot Study
Acronym: ImmersiveAOT
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Siena, Italy (Unknown)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, Professor, IRCCS Fondazione Stella Maris
Other Study IDs: ImmersiveAOT
Record Dates: First submitted 2026-01-16; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); CP (Cerebral Palsy); Motor Imagery; Action Observation
Keywords: Immersive; AOT; Cerebral Palsy; Motor Imagery; haptic gloves; eye-tracker; Mirror Neuron System; EEG; multisensory
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Study Group): 20 participants aged 7-25 years diagnosed with Cerebral Palsy (CP)
- Group 2 (Control Group): 20 participants with typical development (TD) aged 7-25

SUMMARY:
The discovery of the Mirror Neuron System (MNS) has promoted the development of rehabilitation techniques such as Action Observation Treatment (AOT) and Motor Imagery (MI). These are based on the principle that neural circuits active during execution, also activate during the observation or imagination of movements. These techniques have been found to be effective in several clinical populations including children with Cerebral Palsy (CP), the most common childhood-onset motor disorder. We hypothesize that a multimodal version of AOT, integrating not only visual stimuli (standard practice) but also auditory and tactile stimuli, could further enhance the activation of the MNS. In fact, everyday actions naturally involve multiple sensory channels, and evidence indicate that audio-visual action observation activates the MNS more intensely than visual stimuli alone, thus offering a potential improvement for CP rehabilitation.

The primary aim of this observational pilot study, conducted at IRCCS Fondazione Stella Maris, is to verify whether a multisensory (=immersive) AO session - combining visual, auditory, and tactile stimuli - produces greater activation of the MNS, than a traditional session (visual AO alone). Neural correlates will be measured through high-density Electroencephalography (hdEEG), with a specific focus on the modulation of the sensorimotor mu rhythm. Twenty children and adolescents with CP, aged 7-25 years, and 20 typically developing (TD) aged-matched peers will be recruited in the study. The study also aims to assess the level of participants' attention during stimuli presentation through eye tracking, and to verify whether immersive AO can influence MI abilities, measured through specific tasks and questionnaires (i.e., Motor Imagery Questionnaire for Children (MIQ-C, aged 7-12) and the Motor Imagery Questionnaire - 3 (MIQ-3) for adolescent). In an initial phase of the study both questionnaires will be the validated in a separate sample of 120 TD Italian children and 120 Italian adolescents or adults. The absence of intellectual disability will be assessed using the age-appropriate version of Raven's Progressive Matrices test.

Each participant will undergo two EEG sessions: the immersive session will consist of watching first-person videos accompanied by auditory stimuli consistent with the action and tactile stimuli provided by TouchDIVER Pro haptic gloves (Weart, CE-marked device), suitably adapted for the paediatric population. The traditional session will consist of watching videos without sounds or any tactile additional stimulus. The two sessions will be performed in a in random order. In both sessions, after the observation phase, participants will be asked to perform or imagine the same actions presented in the videos. During observation, eye movements and gaze behavior will be monitored using an eye tracking system. Throughout each session, cortical activity will be recorded using a 128-channel hdEEG net. The sessions will be video-recorded to accurately monitor participants motor behavior, response times, and compliance with the protocol.

At the end of each EEG session, participants will be administered the MIQ-C or MIQ-3 questionnaire and a short task to assess MI abilities. In this task, participants will watch some of the videos previously used during the EEG session and will then be asked to imagine the same action. In this case, their imagery will be interrupted at specific time points, and they will be asked to select, from two images, the moment of the action corresponding to the point at which they were interrupted.

Data analysis will examine within- and between-groups differences for the immersive AO vs the traditional AO. Correlation analysis will be also performed between neurophysiological data, attentional data, questionnaires, MI responses and standardized clinical assessments ( for the CP group), in order to understand how the participants' motor and cognitive abilities influence the activation of the circuits involved in the experimental tasks.

ELIGIBILITY:
Study Group: Inclusion Criteria:

* Confirmed diagnosis of cerebral palsy, documented by clinical history and instrumental examinations;
* Age between 7 and 25 years at the time of recruitment;
* At least one verbal or nonverbal intellectual functioning index >= 70, to ensure understanding and compliance with the tasks required.

Exclusion Criteria:

* Severe sensory disorders that compromise the feasibility of the study;
* Neuropsychiatric comorbidity that precludes participation in the study.

Control group: Inclusion Criteria

* Age between 7 and 25 years at the time of recruitment;
* Absence of intellectual disability, assessed through age-appropriate versions of the Raven's Progressive Matrices (Coloured Progressive Matrices for children up to 11 years; Standard Progressive Matrices for participants aged 12 years and older), yielding scores within the normative range and used to estimate non-verbal fluid intelligence;
* Age-appropriate academic performance with no reports of significant learning difficulties, as verified through parental interview;
* Absence of known neurological or psychiatric disorders, confirmed through parental interview;
* Absence of motor impairments, defined as scoring above the 25th percentile on the Movement Assessment Battery for Children, Second Edition (MABC-2).

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: For this study, 20 children, adolescents, and young adults with typical development will be recruited (community sample), toghether with 20 children and adolescents diagnosed with CP (recruit at the IRCCS Fondazione Stella Maris).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological data (hdEEG) | one hour per session
  The primary outcome will be represented by the neurophysiological data obtained from the two recording sessions. Spectral and time-frequency analyses will be performed to examine the reactivity of specific frequency bands (e.g., sensorimotor mu rhythm and attentional alpha rhythm) in relation the presented stimuli. Event-related desynchronization/synchronization (ERD/ERS) patterns will be compared across sessions and between groups.

SECONDARY OUTCOMES:
Attention and motor imagery data | One hour per session
  Secondary outcomes will be represented by data on participants' attention (eye tracker) and MI. Analysis of data obtained from the eye tracking will focus on eye movements, stimulus fixation duration, and saccadic movements during video viewing. Scores from the MIQ-C and MIQ-3 questionnaires and the MI task results will also be included. These data will compared across sessions and between groups. Also, aorrelation analyses with EEG data will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Sgandurra, PhD, MD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Calambrone, Pisa, Italy

REFERENCES:
- [Result] Rizzolatti G, Fadiga L, Gallese V, Fogassi L. Premotor cortex and the recognition of motor actions. Brain Res Cogn Brain Res. 1996 Mar;3(2):131-41. doi: 10.1016/0926-6410(95)00038-0. PMID 8713554
- [Result] Pineda JA. The functional significance of mu rhythms: translating "seeing" and "hearing" into "doing". Brain Res Brain Res Rev. 2005 Dec 1;50(1):57-68. doi: 10.1016/j.brainresrev.2005.04.005. Epub 2005 May 31. PMID 15925412
- [Result] Paulus M, Hunnius S, Bekkering H. Neurocognitive mechanisms underlying social learning in infancy: infants' neural processing of the effects of others' actions. Soc Cogn Affect Neurosci. 2013 Oct;8(7):774-9. doi: 10.1093/scan/nss065. Epub 2012 Jun 11. PMID 22689219
- [Result] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Result] Marshall PJ, Meltzoff AN. Neural mirroring systems: exploring the EEG mu rhythm in human infancy. Dev Cogn Neurosci. 2011 Apr;1(2):110-23. doi: 10.1016/j.dcn.2010.09.001. PMID 21528008
- [Result] Kohler E, Keysers C, Umilta MA, Fogassi L, Gallese V, Rizzolatti G. Hearing sounds, understanding actions: action representation in mirror neurons. Science. 2002 Aug 2;297(5582):846-8. doi: 10.1126/science.1070311. PMID 12161656
- [Result] Keysers C, Kohler E, Umilta MA, Nanetti L, Fogassi L, Gallese V. Audiovisual mirror neurons and action recognition. Exp Brain Res. 2003 Dec;153(4):628-36. doi: 10.1007/s00221-003-1603-5. Epub 2003 Aug 23. PMID 12937876
- [Result] Keysers C, Kaas JH, Gazzola V. Somatosensation in social perception. Nat Rev Neurosci. 2010 Jun;11(6):417-28. doi: 10.1038/nrn2833. Epub 2010 May 6. PMID 20445542
- [Result] Kaplan JT, Iacoboni M. Multimodal action representation in human left ventral premotor cortex. Cogn Process. 2007 Jun;8(2):103-13. doi: 10.1007/s10339-007-0165-z. Epub 2007 May 15. PMID 17503101
- [Result] Hetu S, Gregoire M, Saimpont A, Coll MP, Eugene F, Michon PE, Jackson PL. The neural network of motor imagery: an ALE meta-analysis. Neurosci Biobehav Rev. 2013 Jun;37(5):930-49. doi: 10.1016/j.neubiorev.2013.03.017. Epub 2013 Apr 10. PMID 23583615
- [Result] Fox NA, Bakermans-Kranenburg MJ, Yoo KH, Bowman LC, Cannon EN, Vanderwert RE, Ferrari PF, van IJzendoorn MH. Assessing human mirror activity with EEG mu rhythm: A meta-analysis. Psychol Bull. 2016 Mar;142(3):291-313. doi: 10.1037/bul0000031. Epub 2015 Dec 21. PMID 26689088
- [Result] Demas J, Bourguignon M, Perivier M, De Tiege X, Dinomais M, Van Bogaert P. Mu rhythm: State of the art with special focus on cerebral palsy. Ann Phys Rehabil Med. 2020 Oct;63(5):439-446. doi: 10.1016/j.rehab.2019.06.007. Epub 2019 Jul 9. PMID 31299375
- [Result] Bakker M, Sommerville JA, Gredeback G. Enhanced Neural Processing of Goal-directed Actions After Active Training in 4-Month-Old Infants. J Cogn Neurosci. 2016 Mar;28(3):472-82. doi: 10.1162/jocn_a_00909. Epub 2015 Dec 17. PMID 26679217